CLINICAL TRIAL: NCT02217124
Title: Impact of High Fiber Snacks on Adiposity, Glucose Regulation and Appetite in Children
Brief Title: Impact of High Fiber Snacks on Adiposity, Glucose Regulation and Appetite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Principal Investigator, Dr. Shirin Hooshmand, Assistant Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: S17213
Record Dates: First submitted 2014-08-12; First posted 2014-08-15 (Estimated); Last update posted 2017-08-11 (Actual); Status verified 2017-08

CONDITIONS: Obesity
Keywords: apple; high fiber; body composition; children
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Apple group (Experimental): twenty four participants will be randomly selected for the apple group, in which they will receive 37.5 grams equal to 120kcal of dried apples twice a day for eight weeks. This snack of apples will be eaten once between breakfast and lunch and once between lunch and dinner and both will be consumed with an eight ounce bottle of water.
  Interventions: Other: dried apples
- Muffin control (Placebo Comparator): twenty four participants will be randomly selected to make up the muffin control group, in which one 120kcal muffin control snack will be consumed twice each day for eight weeks. The muffin control will be consumed one between breakfast and lunch and one between lunch and dinner, each snack will be consumed with an eight ounce bottled water.
  Interventions: Other: muffin

INTERVENTIONS:
Other: dried apples — 120 calories
  Arms: Apple group
Other: muffin — 120 calories
  Arms: Muffin control

SUMMARY:
The primary objective of the proposed research is to determine the influence of 8 weeks of twice daily consumption of 120 kcal servings of dried apples or a commonly consumed low fat 120kcal muffin on components of obesity (waist circumference [waist measurement], serum glucose [blood sugar], triglycerides [fats in the blood] and HDL-cholesterol, and blood pressure) as well as antioxidant status, inflammatory markers, nutrient intake in overweight and obese individuals. A total of 48 children aged 10-16 years will be randomly assigned to groups and provided with twice daily 120 kcal servings of either dried apples or muffins for 8 weeks of feeding. Prior to initiating the feeding trial and again after 8 weeks, blood samples will be collected and analyzed. During each visit to the lab, subjects will be weighed in minimal clothing, tested for body composition using dual energy X-ray absorptiometry (DXA), bioelectrical impedance (BIA) and air displacement plethysmography (Bod Pod) and blood pressure, and measured for waist circumference. One 24-hour recall will be performed prior to initiation of the study; one recall will be performed throughout the feeding period, and one at the end of the 8 weeks. Dietary intake of energy, macronutrients, vitamins and minerals will be assessed to determine diet quality. All food records will be analyzed using the Nutritionist Pro (First DataBank) software. The potential benefits of the study include determining the effects of consistent snacking and particular snack foods on metabolism and weight management. There are no major risks to subjects in this study. There are minimal risks when performing venipuncture (blood draws) including bruising, perforation of the vein leading to hematoma under skin, light-headedness or dizziness due to fear of needles, and infection. This study will hopefully allow more understanding and insight into the diet of children and the effect of it on body makeup and blood sugar. It is hypothesized that the twice a day apple snack group will have decreased waist circumference, body adiposity, triglycerides and total cholesterol as well as, increased blood glucose uptake at the end of 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* must be between age 10-16
* must be overweight or obese according to growth charts

Exclusion Criteria:

* regular consumers of apples (one per day)
* supplement users other than multivitamin

Ages: 10 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2014-07; Primary Completion 2016-02 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Change from baseline Body Composition at 8 weeks | baseline, 8 weeks
  Height, Weight, waist circumference, Body Mass Index are all used to asses body composition. Bod pod, BIA, and Dexa are also used to obtain the body composition.

SECONDARY OUTCOMES:
Change from baseline of triglycerides at 8 weeks | baseline, 8 weeks
Change from baseline blood glucose at 8 weeks | baseline, 8 weeks
  Used to examine glucose regulation as effected by the apple group intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Shirin Hooshmand, PhD, Principal Investigator — San Diego State University
Locations (1):
- San Diego State Univeristy, San Diego, California, United States